CLINICAL TRIAL: NCT02842996
Title: A Qualitative Study to Ascertain Patient Reported Experience Measures Following Hip Fracture Surgery in the Elderly
Brief Title: Patient Reported Experience Measures Following Hip Fracture Surgery in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: University of Birmingham
Record Dates: First submitted 2016-04-07; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Hip Fractures; Elderly; Emergency Surgery
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient and carer study group: Patients having undergone hip fracture surgery and their care givers.

SUMMARY:
With an ageing population, hip fractures are likely to become a significant public health burden. Hip fracture surgery is associated with significant morbidity and mortality. Patient outcomes and experience underpin the National Health Service (NHS) Constitution in driving quality improvement and performance.

We aim to conduct a qualitative research study to ascertain the important patient and carer reported experience measures following hip fracture surgery in the elderly to improve quality of care and service provision.

To learn about patient and care-giver experience to ascertain which aspects are important to patients and what can be improved.

DETAILED DESCRIPTION:
Rationale for research:

Recovery following hip fracture surgery has been associated with poor functional outcome; (Marcantonio et al. 2001; Luger et al. 2010) these patients may require longer hospital stays, are more often discharged to long-term care, and have a generally poor prognosis for returning home or regaining function in activities of daily living (ADL). (Dolan et al. 2000) Loss to living independently in the community has a significant detrimental effect on their quality of life and some patients have reported that they would rather be dead than experience the loss of independence that results from a hip fracture. (Salkeld et al. 2000) Patients report that going home following hip fracture surgery would be their main priority. (Robinson et al. 2015) Recovery for patients is multi-faceted and includes physical, social and emotional domains. (Miller & Mythen 2014) Increasingly focus is being modified to include patient related experience of the healthcare pathway to inform policymakers, health regulation and service improvement. (Gibbons & Fitzpatrick 2012) Patient public involvement (PPI) via the Clinical Research Ambassador Group (CRAG) at Heart of England NHS Foundation Trust has helped to identify the research question with particular focus on the improving the perioperative care pathway. Members of the CRAG group have reported the impact of hip fracture to include loss of functional ability leading to additional stress for family members. They have advocated a qualitative study to assess the impact on patients and their carers based on their personal experiences. We aim to conduct interviews to ascertain important and relevant patient reported experience measures in elderly patients undergoing hip fracture surgery.

Aims:

To review and evaluate the literature to ascertain the themes related to patient and carer experiences following hip fracture surgery which can improve quality of care.

To conduct interviews to ascertain what are the patient and carer experiences surrounding discharge from hospital following hip fracture surgery? To identify important themes to guide us in improving the care-pathway surrounding patient discharge following fractured neck of femur surgery in the elderly.

To pilot a resource/information pack designed specifically to improve patient and carer experience following hip fracture surgery?

Research questions:

In the published literature what are the themes related to patient and carer experiences following hip fracture surgery which can improve quality of care? What are the patient and carer experiences surrounding discharge from hospital following hip fracture surgery? From patient and carer experience following hip fracture surgery what are the important themes that can improve the discharge pathway for patients and their carers.

What information should be included in a resource pack designed to help patient and carer following hip fracture surgery? Will a resource/information pack designed specifically help to improve patient and carer experience following hip fracture surgery?

Qualitative Interviews:

To explore physical, mental and emotional impact on patient and care-givers following hip fracture surgery we will conduct semi-structured interviews of patients and their care-givers. Participants will include patients who have undergone hip fracture surgery and their named care-giver. Participants will be screened at a single study site using clinical databases as well as reviewing new patients that are admitted on the orthopaedic ward. Patients will be excluded if they are unable to consent or unable to partake in the interview due to speech and language impairment.

Conduct of Interviews:

Semi-structured interviews will be conducted with patients and their carers at their location of choice. This will be at their residence or at the study site; if they choose to travel to the study site their travel expenses will be re-imbursed. If patients and their carers are being interviewed at the same time, we will aim to interview them separately, unless they request to be interviewed together. The interviews will be carried out by one member of the research team this will aim to ensure consistency of interview questions and technique throughout the study. Prior to starting the interview with the participants we will reconfirm consent. The interviews will be audio-recorded and written notes will also be taken.

Ethical considerations and consent:

Written consent will be obtained from participants during their in-patient hospital stay. An informal capacity/consent process will be used by a trained member of the research team. Written and verbal information will be provided about the study, using a suitable style and format for the participant. The researcher will ask the participant to recall study information to check understanding; this together with the clinical teams view will be used to assess capacity to consent. Consent will be sought for:

* Accessing medical records for the purpose of collecting relevant patient outcomes and patient health service use.
* Participating in a face to face interview following hospital discharge. If a patient is deemed to not have capacity they will not be included in the study.

Risks, burdens and benefits:

There is a small risk of distress for the patient and/or their carer during the interview when describing their memories and experiences. There may also be a time-burden to patients and their carers by taking part in the interview. To minimise these factors we will ensure that interviews are conducted on a day and time convenient to the patient and their carer. They will be able to stop the interview at any time and take a break if they require. If the patient/carer request or are identified as requiring support we will offer to contact their general practitioner (GP) on their behalf. The patient and their carer will be interviewed separately but if either requires support or feel vulnerable if left alone they will be interviewed together. If the patient requires the interview to be conducted in the community or at the patient's home there is a risk of the researcher, conducting the interview, to be put in a potential vulnerable situation. This will be minimised by ensuring the researcher follows Birmingham Heartlands Hospital lone worker policy.

Data analysis:

Interviews will be recorded and analysed anonymously with only the author knowing participant details. Data will be transcribed verbatim; transcripts will thereafter be reviewed to check for accuracy. Coding of the transcripts will occur, a second reviewer will check these. Results from the data analysis will guide development of a resource/information pack designed specifically help to improve patient and carer experience following hip fracture surgery.

Dissemination of results:

This study will not directly benefit the participants but it will improve services for patients in the future undergoing hip fracture surgery. It will identify areas of need/support to guide National Health Service (NHS) policymakers and healthcare provision and development of services to facilitate discharge to the community. By understanding the important patient reported experience measures we can go on to use these and compare quality of healthcare in this group of patients to improve care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over.
* Due to have surgical fixation for proximal femoral fracture.
* Care-giver of a patient having undergone surgical fixation for proximal femoral fracture.

Exclusion Criteria:

* Patients admitted with multiple trauma.
* Patients who are unable to speak sufficient English to participate in the interview.
* Patients who are unable to consent due to lack of capacity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged over 65 years undergoing hip fracture surgery. Care-givers of patients having undergone hip fracture surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Patient experiences following hip fracture surgery | 6 months
  Patients views and perceptions around their experience of hip fracture surgery with particular focus surrounding the discharge pathway.
Carer experiences following hip fracture surgery | 6 months
  The views and perceptions of supporting a relative/friend having undergone hip fracture surgery, with particular focus on the discharge pathway.

IPD SHARING:
Plan to Share IPD: No